CLINICAL TRIAL: NCT01554020
Title: Effect of Blood Sugar Take Care on Glucose Metabolism, Determinants of Metabolic Syndrome, and Quality of Life in Prediabetic Adults: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Blood Sugar Take Care and Glucose Metabolism
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change of CRO
Sponsor: NewChapter, Inc. (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 120216-SUS-NWC-BSS-GP
Record Dates: First submitted 2012-03-07; First posted 2012-03-14 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Prediabetes
Keywords: Blood glucose; Insulin sensitivity; Oral glucose tolerance
MeSH Terms: conditions — Prediabetic State; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiherb product (Active Comparator): Herbal product
  Interventions: Dietary Supplement: Blood Sugar Take Care
- Placebo (Placebo Comparator): Maltodextrin control
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blood Sugar Take Care — One 1200 mg soft gel capsule administered 3X/day for duration of study
  Other Names: BSTC
  Arms: Multiherb product
Dietary Supplement: Placebo — One 1200 mg soft-gel capsule administered 3X/day for duration of study
  Arms: Placebo

SUMMARY:
This prospective international clinical trial is a two-arm, double-blind, randomized, placebo-controlled, parallel-group, multicenter study. 112 prediabetic subjects will be randomized to Blood Sugar Take Care or placebo. Randomization will be stratified by gender. The intervention period is 12 weeks. The primary outcome is fasting glucose levels.

ELIGIBILITY:
SUBJECT INCLUSION CRITERIA: STEP 1

1. Age ≥ 18 years
2. Subject meets American Diabetes Association criteria for diabetes testing in asymptomatic, undiagnosed individuals:

   1. If age ≥45 years, subject must have a body mass index ≥ 25 kg/m2 for United States and ≥ 24 kg/m2 for Indonesia
   2. If age <45 years, subject must have a body mass index ≥ 25 kg/m2 for United States and ≥ 24 kg/m2 for Indonesia AND present with at least one of the following risk factors:

      * Have a first-degree relative with diabetes
      * Habitually physically inactive
      * Race is African-American, Hispanic American, Native American, Asian American, or Pacific Islander
      * Have delivered a baby weighing >9 lb or have been diagnosed with gestational diabetes mellitus
      * Hypertensive (≥140/90)
      * Known HDL cholesterol level 35 mg/dl
      * Known triglyceride level ≥250 mg/dl
      * On previous testing, had impaired glucose tolerance or impaired fasting glucose
      * History of vascular disease
3. Stable body weight (<5% change) in the last 3 months
4. Agree to use contraception throughout study period, unless postmenopausal or surgically sterile (females only)
5. Able to understand the nature and purpose of the study including potential risks and side effects
6. Willing to consent to study participation and to comply with study requirements

SUBJECT EXCLUSION CRITERIA

1. Known diabetes (type I or II)
2. Recent use (within 2 weeks of screening) of any dietary supplement including vitamin and mineral complexes; herbal supplements; fish oil; fiber supplements; or any herbal ingredient/product that significantly affects glucose or lipid metabolism
3. Recent use (within 4 weeks of screening) of any prescription or OTC medication that significantly affects glucose or lipid metabolism, including but not limited to, sulfonylureas, meglitinides, biguanides, thiazolidinediones, alpha-glucosidase inhibitors, DPP-4 inhibitors, systemic corticosteroids, statins, fibrates, niacin, and bile acid sequestrants
4. Daily use of nonsteroidal anti-inflammatory drugs (NSAIDS); (daily baby aspirin use acceptable)
5. Any comorbidity that could, in the opinion of the investigator, preclude the subject's ability to successfully and safely complete the study or that may confound study outcomes
6. Anticipated changes in dietary patterns or physical activity levels during the study, including attempts at body weight reduction
7. Eating disorder
8. Polycystic ovary syndrome
9. Known allergies to any substance in the study product
10. Pregnant or breastfeeding women
11. History of alcohol, drug, or medication abuse
12. Participation in another study with any investigational product within 3 months of screening
13. Recent (<3 months) gastrointestinal surgery or any planned surgery during the treatment period

SUBJECT INCLUSION CRITERIA: STEP 2

1. Fasting glucose between 95 and 130 mg/dl, based on portable glucometer reading

SUBJECT INCLUSION CRITERIA: STEP 3

1. Impaired fasting glucose, based on the American Diabetes Association definition of fasting serum glucose between 100 and 125 mg/dl
2. Impaired glucose tolerance, based on the American Diabetes Association definition of serum glucose between 140 and 199 mg/dl 2 hours after a 75 g glucose load

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose | 12 weeks

SECONDARY OUTCOMES:
Insulin sensitivity index | 12 weeks
Fasting insulin | 12 weeks
Homeostasis Model Assessment of Insulin Resistance | 12 weeks
Quantitative insulin sensitivity check index | 12 weeks
Insulin secretion/insulin resistance index | 12 weeks
Glycosylated hemoglobin (HbA1c) | 12 weeks
High-sensitivity C-reactive protein | 12 weeks
High-molecular weight adiponectin | 12 weeks
Lipids (total cholesterol, HDL, LDL, VLDL, triglycerides) | 12 weeks
Body composition | 12 weeks
  height/weight, body mass index, waist circumference, hip circumference, waist-to-hip ratio
WHO Quality of Life Questionnaire | 12 weeks
Comprehensive metabolic panel | 12 weeks
Complete blood count | 12 weeks
Adverse events | 12 weeks
Gastrointestinal Symptom Rating Scale | 12 weeks
Pulse | 12 weeks
Blood pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Larry Miller, PhD, Principal Investigator — Sprim Advanced Life Sciences
Locations (1):
- SPRIM, San Francisco, California, United States